CLINICAL TRIAL: NCT06734338
Title: Validation of the STUMBL Score for Risk Stratification in Emergency Department Patients With Blunt Thoracic Trauma: A Prospective Observational Study in Iraq
Brief Title: Validation of the STUMBL Score for Blunt Thoracic Trauma
Acronym: STUMBL
Status: Not yet recruiting | Type: Observational
Sponsor: Al-Nahrain University (Other)
Responsible Party: Principal Investigator, Abdul-Ilah R. Khamis, Principal Investigator, Al-Nahrain University
Other Study IDs: UNCOMIRB20241212; 012 (Other: Nahrain Medical Research Collective (NMRC))
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Chest Trauma
Keywords: STUMBL; Trauma; Chest
MeSH Terms: conditions — Thoracic Injuries; Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This prospective observational study aims to validate the STUMBL score for risk stratification in emergency department patients with blunt thoracic trauma in Iraq. The main questions it seeks to answer are:

How accurately does the STUMBL score predict mortality and critical outcomes such as ICU admission or advanced interventions? How well does the score stratify patients by injury severity in a resource-limited setting? Are there demographic or clinical factors that influence the score's predictive performance?

Participants will:

Be assessed using the STUMBL score upon arrival at the emergency department to predict risk levels.

Have demographic and clinical data, including age, gender, injury mechanism, comorbidities, and length of hospital stay, collected to explore potential associations with outcomes.

DETAILED DESCRIPTION:
Blunt thoracic trauma (BTT) is a significant cause of morbidity and mortality in emergency department (ED) patients worldwide. The complexity of BTT management arises from the diverse range of injuries that can occur, including rib fractures, pneumothorax, and hemothorax, which can lead to life-threatening complications if not promptly identified and treated. Studies indicate that the rise in mortality and long-term morbidity can be clearly linked to the number of rib fractures sustained. Road traffic collisions are the predominant cause of major blunt injury. BTT is more common, with relative incidence being estimated at 72-83.5% versus penetrating trauma at 16.5-28%. In emergency settings, timely and accurate assessment of patients with blunt thoracic injuries is crucial for optimizing outcomes. Thereby, there is a need for valid systems that can be effectively utilized in emergency departments to enhance clinical decision-making in a short-term manner.

The STUMBL (STUdy of the Management of BLunt chest wall trauma) score was developed to assist in clinical decision-making for patients with blunt chest wall trauma. This model includes five risk factors: patient age, the number of rib fractures, chronic lung disease, pre-injury use of anticoagulants, and oxygen saturation levels. Unlike other scoring systems that focus solely on anatomical variables and age, the STUMBL score uniquely incorporates clinical variables such as chronic lung disease and anticoagulation. A huge benefit of the STUMBL score is that these variables are all routinely measured in the ED. The score has reached a sensitivity of 80%, a specificity of 96%, a positive predictive value (PPV) of 93%, and a negative predictive value (NPV) of 86% for predicting complications following blunt chest wall trauma. By integrating essential clinical parameters, the STUMBL score helps clinicians identify patients at high risk for adverse outcomes. Each patient is evaluated based on several risk factors. A final risk score of ≥11 indicates a significant risk of developing complications, and a total risk score exceeding 25 is considered sufficiently high to require admission to the intensive care unit (ICU).

The STUMBL score has shown potential across various healthcare settings. However, its validation in varied populations, especially in low-resource areas, remains limited. In the context of Iraqi EDs, the applicability of the STUMBL score has not been thoroughly investigated. As healthcare systems face challenges related to resource, training, and infrastructure limitations, the integration of evidence-based tools like the STUMBL score could significantly improve patient care. The burden of trauma is compounded by ongoing conflict and limited healthcare resources, leading to an urgent need for effective trauma management protocols. This study aims to evaluate the performance of the STUMBL score among ED patients presenting with blunt thoracic trauma in Iraq.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with blunt thoracic trauma (e.g., motor vehicle accidents, falls, or direct impacts to the chest).
* Patients who present within 4 hours of sustaining the injury.
* Patients or their legal guardians must provide informed consent to participate in the study.

Exclusion Criteria:

* Patients with penetrating chest trauma (e.g., stab wounds, gunshot wounds).
* Patients with other life-threatening injuries that overshadow the thoracic trauma (e.g., head or abdominal trauma).
* Pregnant women due to potential risks related to radiation or certain diagnostic procedures.
* Pediatric patients under 18 years of age.
* Patients with a history of major thoracic surgery (e.g., prior lung or heart surgery) that may interfere with the assessment of trauma severity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adult patients (18 years and older) presenting to the emergency department at Al-Kadhimiya Teaching Hospital, Baghdad, with blunt thoracic trauma. Participants will be assessed based on injury mechanisms such as motor vehicle accidents, falls, or direct impacts, along with the severity of the trauma. Both male and female patients, regardless of comorbidities, will be included to evaluate the STUMBL score's applicability across different demographics and clinical profiles.
Sampling Method: Non-Probability Sample
Enrollment: 188 (Estimated)
Dates: Start 2025-04-20 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2025-07-20 (Estimated)

PRIMARY OUTCOMES:
In hospital mortality | In-Hospital Phase (average of 10 days through discharge); Post-Discharge Follow-Up: Day 7, Day 30
  Mortality (death) during hospitalization.
Accuracy Assessment of the STUMBL score | the first 4 hours after ER admission
  The score ranges from 1 to 30. ≥11 is particularly significant, as it indicates a higher risk of complications.

SECONDARY OUTCOMES:
Length of Hospitalization | Up to discharge, an average of 10 days
  The total duration of a patient's stay in the hospital, measured from the date of admission to the date of discharge. This includes all days spent in general wards, intensive care units (ICU), and other hospital departments as part of their treatment course.
Rate of ICU Admission | Up to discharge, an average of 10 days
  The requirement for admission to the intensive care unit (ICU) is determined by the presence of severe clinical deterioration, significant complications, or the need for advanced monitoring and life-support measures.
Rate of Participants Requiring Surgical Intervention | Up to discharge, an average of 10 days
  need for surgical intervention during a trauma patient's hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Yaser aamer Eisa Alhaibi, Assistant professor, Study Director — College Of Medicine - Nahrain University
Locations (1):
- College of Medicine - Al-Nahrain University, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelderman I, Dickhoff C, Bloemers FW, Zuidema WP. Very long-term effects of conservatively treated blunt thoracic trauma: A retrospective analysis. Injury. 2024 Apr;55(4):111460. doi: 10.1016/j.injury.2024.111460. Epub 2024 Mar 2. PMID 38458000
- [Background] Mistry RN, Moore JE. Management of blunt thoracic trauma. BJA Educ. 2022 Nov;22(11):432-439. doi: 10.1016/j.bjae.2022.08.002. Epub 2022 Oct 1. No abstract available. PMID 36304913
- [Result] Mukerji S, Tan E, May C, Micanovic C, Blakemore P, Phelps K, Melville H, Jones P. Retrospective validation of a risk stratification tool developed for the management of patients with blunt chest trauma (the STUMBL score). Emerg Med Australas. 2021 Oct;33(5):841-847. doi: 10.1111/1742-6723.13740. Epub 2021 Feb 17. PMID 33599054
- [Result] Callisto E, Costantino G, Tabner A, Kerslake D, Reed MJ. The clinical effectiveness of the STUMBL score for the management of ED patients with blunt chest trauma compared to clinical evaluation alone. Intern Emerg Med. 2022 Sep;17(6):1785-1793. doi: 10.1007/s11739-022-03001-0. Epub 2022 Jun 23. PMID 35739456
- [Result] Battle C, Cole E, Whelan R, Baker E. Scoping review of the literature to ascertain how the STUMBL Score clinical prediction model is used to manage patients with blunt chest wall trauma in emergency care. Injury. 2023 Jul;54(7):110796. doi: 10.1016/j.injury.2023.05.027. Epub 2023 May 7. PMID 37208252
- [Result] Battle C, Cole E, Carter K, Baker E. Clinical prediction models for the management of blunt chest trauma in the emergency department: a systematic review. BMC Emerg Med. 2024 Oct 12;24(1):189. doi: 10.1186/s12873-024-01107-6. PMID 39395934